CLINICAL TRIAL: NCT01891435
Title: A Randomized Controlled Clinical Trial on the Antipyretic Efficacy of Oral Paracetamol, Intravenous Paracetamol and Intramuscular Diclofenac in Patients Presenting With Fever to Emergency Department
Brief Title: The Antipyretic Efficacy of Oral and Intravenous Paracetamol and Intramuscular Diclofenac in Patients Presenting With Fever.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Firjeeth C Paramba, Specialist, Emergency Department, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9070/09
Record Dates: First submitted 2013-06-21; First posted 2013-07-03 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-06

CONDITIONS: Fever; Reduction in Temperature
Keywords: antipyretics; oral paracetamol; intravenous paracetamol; intramuscular diclofenac; emergency department
MeSH Terms: conditions — Fever; Emergencies | interventions — Acetaminophen

ARMS (3):
- oral paracetamol (Active Comparator): patients in this arm will receive 1000mg of oral paracetamol
  Interventions: Drug: Oral paracetamol
- Intravenous paracetamol (Active Comparator): patients in this arm will receive 1000 mg of intravenous paracetamol
  Interventions: Drug: Intravenous paracetamol
- Intramuscular Diclofenac (Active Comparator): patients in this arm will receive 75 mg of intramuscular diclofenac sodium
  Interventions: Drug: Intramuscular diclofenac

INTERVENTIONS:
Drug: Oral paracetamol — after giving medicine temperature is checked every 30 minutes for 2 hours
  Arms: oral paracetamol
Drug: Intravenous paracetamol — after giving medicine temperature is checked every 30 minutes for 2 hours
  Arms: Intravenous paracetamol
Drug: Intramuscular diclofenac — after giving medicine temperature is checked every 30 minutes for 2 hours
  Arms: Intramuscular Diclofenac

SUMMARY:
A randomized clinical trial to check the antipyretic efficacy of oral and intravenous paracetamol and intramuscular diclofenac sodium in patients presenting with fever to emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the age of 14-75 years with an oral temperature of more than 38.5 C

Exclusion Criteria:

* History of allergy to any of the drugs in the study
* Had taken antipyretics within 8 hours
* Renal, hepatic or haematological disorders
* bronchial asthma, peptic ulcer disease, vomiting
* Pregnant or lactating women

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Reduction in temperature in every thirty minutes till 120 minutes after receiving antipyretics | Reduction in temperature is checked every 30 minutes for a maximum of 120 minutes
  Once the patients fulfill the inclusion criteria, they are randomly assigned to receive one of the three medications in the study ( oral paracetamol, intravenous paracetamol or intramuscular diclofenac). Baseline temperature is recorded using a standard thermometer. Then reduction in temperature is recorded every 30 minutes for 2 hours.

CONTACTS AND LOCATIONS:
Overall Officials: osama H Mohammed, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad medical corporation, Doha, Qatar